CLINICAL TRIAL: NCT05655507
Title: A Phase 1, Study to Evaluate the Pharmacokinetics and Safety of Zuranolone in Adolescents (12 to 17 Years of Age) With Major Depressive Disorder
Brief Title: Zuranolone Pharmacokinetics (PK) and Safety Study Adolescent Participants With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 217-CLP-118; NCT05655507 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression; Pediatrics; Child; Adolescent; SAGE-217; Zuranolone
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — zuranolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zuranolone (Experimental): Participants will be enrolled to receive Zuranolone orally, during the daytime on Day 1 and in the evening on Days 2 to 14. The first 10 enrolled participants will receive 50 mg (participants with a body weight of 54 kg or greater) or 40 mg (participants with a body weight less than 54 kg) once daily. The remaining participants will receive 40 mg once daily with the opportunity to down titrate to 30 mg if 40 mg is not tolerated.
  Interventions: Drug: Zuranolone

INTERVENTIONS:
Drug: Zuranolone — Administered as capsules
  Other Names: SAGE-217, BIIB125

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics and safety of Zuranolone in adolescents (ages 12 to 17 years) with MDD.

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In December 2024, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime DSM-5 (KSADS-PL DSM-5) criteria for MDD.
* Participant has a Children's Depression Rating Scale-Revised (CDRS-R) total score greater than or equal to 40 at screening and Day 1.
* Participant's parent/caregiver is able to attend all scheduled study visits, oversee administration of study drug and complete assessments per the protocol.
* Participant has a body weight greater than or equal to 20 kg and a body mass index greater than fifth percentile and less than ninety-fifth percentile for age at Screening.
* Participant is a post-pubertal (has experienced menarche) female (sex assigned at birth), 12 to 17 years of age, inclusive, at the time informed consent/assent is obtained.

Exclusion Criteria:

* Participant has a history of psychosis, bipolar disorder, autism, seizures, or other restricted comorbid psychiatric or neurological conditions and has treatment-resistant depression.
* Participant has a known diagnosis of intellectual disability or is unable to communicate with the study investigator or research team.
* Participant has a history of suicidal behavior or is currently at risk of suicide in the opinion of the investigator.
* Participant has a recent history of Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM 5) alcohol or drug use disorder or has clinically significant alcohol or drug misuse as judged by the investigator.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of Zuranolone | At multiple timepoints post dose on Days 1, 8 and 15
  PK Parameters of Zuranolone will be assessed.

SECONDARY OUTCOMES:
Percentage of Participants With at Least one Treatment Emergent Adverse Event (TEAE) | Up to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (4):
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/